CLINICAL TRIAL: NCT05391490
Title: Allogeneic T Cells Expressing T Cell Receptor-KDEL and the Chimeric Antigen Receptor CAT19 for the Treatment of Advanced CD19+ Malignancies
Acronym: KCAT19
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/126900; 2021-002878-88 (EudraCT Number)
Record Dates: First submitted 2022-05-16; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Blood Cancer
Keywords: CAR T cells; leukemia; lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma

STUDY DESIGN:
Intervention Model Description: Single-centre, non-randomised, open-label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product (ATIMP)
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Trial (Experimental): Treatment with Lymphodepletion followed by a dose of KCAT19 T cells.
  Interventions: Genetic: KCAT19 T cells

INTERVENTIONS:
Genetic: KCAT19 T cells — Allogeneic, cord unit derived KCAT19 T cells

SUMMARY:
KCAT19 is a single-centre, non-randomised, open-label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product (ATIMP) in adults (age 16-65 years) with high risk, relapsed/refractory (r/r) B cell malignancies.

DETAILED DESCRIPTION:
The aims of this study are to make sure these KCAT19 T cells can be made in the lab, assess if these therapies are safe and also obtain some initial information that these CAR T cells work in patients with B-cell malignancies.

Following patent's informed consent and registration into the trial, allogeneic HLA-matched cord blood donor T cells will be couriered to the Centre for Cell, Gene & Tissue Therapeutics (CCGTT) at the Royal Free Hospital (RFH) where the KCAT19 T cells will be manufactured. The first 3 patients treated on KCAT19 will be HLA matched 4-6/6 with a cord-blood donor and the remaining patients registered will be HLA matched 0-6/6 if confirmed by the IDMC.

KCAT19 T cells are classified as advanced therapy investigational medicinal products (ATIMPs) and manufacture will take approximately 15 days.

Briefly, the allogeneic cord-blood derived T cells are grown in the presence of a lentivirus which transfers specific genes into the T cells (part of the white blood cells). The genes enable the T cells to express a protein which can recognise a target protein (CD19) present on the surface of the malignant B-cells and attack them. The genetically modified cells are tested to ensure they comply with the specified quality release criteria and frozen at RFH. The ATIMPs are couriered to the trial site with a special shipper (maintaining temperature below -130C) to be administered to the patient when needed. During the ATIMP manufacturing period, patients may receive "holding" chemotherapy or immunotherapy as per institutional practice to maintain disease control. Prior to infusion of the KCAT19 T cells, patients will be admitted to hospital to have pre-conditioning therapy with 2 anticancer drugs: cyclophosphamide and fludarabine.

Patients will then receive the KCAT19 T cell infusion on day 0. The KCAT19 T cells are given as an intravenous infusion. Patients will be closely monitored at the participating trial site for a minimum of 14 days after the KCAT19 T cells infusion with regular observations and blood tests (detailed in the protocol) to assess for potential toxicities. Disease assessment will take place at; baseline, month 1, month 6 and month 12 post-KCAT19 T cell infusion.

Following discharge, patients will be followed up monthly for the first 6 months, then 6 weekly until 12 months post KCAT19 T infusion, followed by quarterly visits for a further year before annual visits until the end of the trial is declared (Year 3 - Year 10).

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-65 years
2. Relapsed or refractory B cell malignancy following at least 2 prior lines of therapy:

   B-ALL: relapsed or refractory B-ALL following standard therapy, requiring salvage, in whom alternative therapies are deemed inappropriate by their treating physician Or LBCL: relapsed/refractory DLBCL (incl. transformed FL but not Richter's transformation) or PMBCL following ≥2 prior lines of therapy which must include Rituximab, anthracycline and autologous CD19 CAR, (unless CD19 CAR cannot be manufactured) Or MCL: relapsed/ refractory disease following ≥2 lines of therapy which must include Rituximab, Bruton's tyrosine kinase inhibitor and autologous CD19CAR therapy (unless CD19 CAR cannot be manufactured) Or Indolent B-NHL (either Follicular Lymphoma, Marginal Zone Lymphoma or other low-grade lymphoma) which is relapsed / refractory following ≥2 prior lines of therapy which must include anti-CD20 therapy and chemotherapy with anthracycline or bendamustine.
3. CD19+ disease
4. Agreement to have a pregnancy test, use adequate contraception (if applicable)
5. Written informed consent

Exclusion Criteria:

1. CD19 negative disease
2. Active CNS involvement of disease
3. Diagnosis of chronic lymphocytic leukaemia/ small lymphocytic lymphoma or Burkitt lymphoma
4. Active hepatitis B, C or HIV infection
5. Oxygen saturation ≤ 90% on air
6. Bilirubin >2 x upper limit of normal
7. GFR <30ml/min
8. Women who are pregnant or breast feeding
9. Stem Cell Transplant patients only: active significant acute GvHD (overall Grade ≥ II, Modified Glucksberg criteria) or moderate/severe chronic GvHD (NIH consensus criteria) requiring immunosuppressive therapy and/or systemic steroids
10. Karnofsky score <60%
11. Known allergy to albumin or DMSO
12. Patients receiving corticosteroids at a dose of >5 mg prednisolone per day (or equivalent) that cannot be discontinued
13. Life expectancy <3 months
14. Cardiac dysrhythmias (excluding well-controlled AF or other supraventricular tachycardia) or significant cardiac disease and left ventricular ejection fraction <40%
15. Patients who can reasonably access autologous CD19 CAR treatment as part of standard of care or a clinical trial*

    * These patients will be initially considered for autologous treatment in preference to enrolling on KCAT19

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2034-11 (Estimated)

PRIMARY OUTCOMES:
KCAT 19 T cell generation feasibility | Up to 28 days after last patient is recruited
  Feasibility of generation of T cell receptor-negative KCAT19 T cells as evaluated by the number of therapeutic products generated.
KCAT19 T cell Toxicity | Up to 28 days after last patient treated
  Toxicity following KCAT19 T cell administration as evaluated by the incidence of grade 3-5 toxicity causally related to the ATIMP

SECONDARY OUTCOMES:
Response rate | 6 months after last patient treated with ATIMP
  Proportion of responders and depth of response at 1 and 6 months post ATIMP infusion
KCAT19 T cell persistence | After last treated patient completes the 2 year follow up visit
  Persistence and frequency of circulating KCAT19 T cells in peripheral blood as assessed by flow cytometry
KCAT19 T cell persistence | After last treated patient completes the 2 year follow up visit
  Persistence and frequency of circulating KCAT19 T cells in peripheral blood as assessed by qPCR
Hypogammaglobulinaemia and B cell aplasia | 2 years after last patient treated
  Incidence and duration of hypogammaglobulinaemia and B cell aplasia
Time to Disease Progression | 2 years after last patient treated
  Time to Disease Progression
Event-Free survival | 2 years after last patient treated
  Event-Free Survival at 1 and 2 years after immunotherapy with KCAT19 T cells
Overall Survival | 2 years after last patient treated
  Overall survival at 1 and 2 years after immunotherapy with KCAT19 T cells

IPD SHARING:
Plan to Share IPD: No